CLINICAL TRIAL: NCT04958057
Title: Social Risks-Focused Lifestyle Intervention to Reduce Preeclampsia in AA Women
Brief Title: Social Risks-Focused Lifestyle Intervention to Reduce Preeclampsia (SAIL)
Acronym: SAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Anna Palatnik, MD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO00041206; 847482 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2021-06-28; First posted 2021-07-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Group prenatal care with a focus on preeclampsia prevention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine prenatal care (No Intervention): Routine prenatal care: All women participating in the study will receive routine prenatal care by their obstetric provider, consisting of 1 prenatal visit a month up to 28 weeks of gestation, 1 prenatal visit every 2 weeks during 28-36 weeks and weekly visits during 36-40 weeks.
- SAIL intervention (Experimental): 6 monthly group sessions with the study nurse with a background in prenatal care and the PI that will include each group will include preeclampsia education, coaching on stress management, resource navigation, and training in problem solving.
  Interventions: Behavioral: SAIL

INTERVENTIONS:
Behavioral: SAIL — 6 monthly group sessions with the study nurse with a background in prenatal care and the PI that will include each group will include preeclampsia education, coaching on stress management, resource navigation, and training in problem solving.
  Other Names: SociAl rIsks-focused Lifestyle intervention
  Arms: SAIL intervention

SUMMARY:
Preeclampsia is a disease of pregnancy and first few weeks after birth. It is diagnosed as new onset of high blood pressure and injury to organs such as kidneys, liver, and brain. Preeclampsia is growing at a rapid rate - rate that exceeds diabetes and heart disease. Over half a million lives lost each year to preeclampsia. Women with a history of preeclampsia have 3-4 times the risk of high blood pressure. They also have double the risk for heart disease and stroke. Racial and ethnic disparities are present in preeclampsia. Black women are at higher risk of developing preeclampsia. They are also at much higher risk of dying from preeclampsia than other women. The reasons behind such disparities are unclear. What may explain these differences are social determinants of health. The contribution of social determinants to differences in preeclampsia is well recognized. However, a major gap in research remains strategies that address these factors. Our study will test a lifestyle intervention incorporating social risk factors to reduce the risk of preeclampsia.

DETAILED DESCRIPTION:
Preeclampsia is a significant global health problem affecting over 10 million pregnancies each year. Preeclampsia disproportionately burdens ethnic minority women, especially African American women when compared to non-Hispanic white women. Once diagnosed with preeclampsia, African women are 3 times more likely to die of preeclampsia compared to their white counterparts. Evidence supports contribution of social risk factors towards racial and ethnic disparities seen with preeclampsia. However, currently, there are few trials that examine efficacy of social risks-focused lifestyle interventions on reduction of preeclampsia and its complications. This proposal is designed to address this crucial gap by testing feasibility (Aim 1), acceptability (Aim 1) and efficacy (Aim 2) of a social risks-focused lifestyle intervention to reduce preeclampsia in pregnant inner-city African American women. The intervention will be delivered via a randomized control trial design (N=100), with 6 monthly group sessions conducted in the second and third trimesters. The overall hypothesis is that the intervention will be feasible and acceptable, and that women randomized to the intervention group will have lower blood pressure and lower rates of preeclampsia compared with women receiving routine prenatal care.

ELIGIBILITY:
Inclusion Criteria:

* self-report as African-American/Non-Hispanic black
* residence in inner-city Milwaukee
* nulliparity
* gestational age at enrollment <=16 weeks
* able and willing to give informed consent

Exclusion Criteria:

* not able to communicate in English
* major fetal anomaly
* psychiatric illness that precludes group participation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Retention | Post intervention measured at the completion of the last study visit, 3 years
  Retention will be measured by session attendance rates.
Systolic and diastolic blood pressure: Post Intervention | Post intervention/at the last study visit, up to 40 weeks
  BP will be taken by a study trained and certified research assistant using the study OMRON automated device.
Systolic and diastolic blood pressure: 6 Weeks Postpartum | At 6 weeks postpartum visit
  BP will be taken by a study trained and certified research assistant using the study OMRON automated device.

SECONDARY OUTCOMES:
Preeclampsia | At the 6 weeks postpartum visit through patient interview, confirmed with medical record review
  The rate of preeclampsia diagnosis will be compared between intervention and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
The proposed study will be conducted, and the data analyzed, and results disseminated in an objective and transparent manner. All investigators are aware of and agree to abide by the principles for sharing research resources, as described by NIH in "Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Programs."